Clinical Study Report: 20140254 Primary Analysis


# 16.1.9 Documentation of Statistical Methods



Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


## STATISTICAL ANALYSIS PLAN

Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of AMG 334 on Exercise Time During a Treadmill Test in Subjects With Stable Angina

**AMG 334** 

Protocol Number: 20140254

Version: Version 2.0

Date: 07 January 2017

Authors:

NCT Number: 2575833
This NCT number has been applied to the document for purposes of posting on clinicaltrials.gov

**AMGEN®** 




Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017 Page 2

## **Table of Contents**

| Table | of Abb | previations4 |
|---|---|---|
| 1. | Introdu | ıction5 |
| 2. | Objecti<br>2.1<br>2.2<br>2.3 | ives 5 Primary 5 Secondary 5 Safety 5 |
| 3. | Study (<br>3.1<br>3.2 | Overview5Study Design5Sample Size5 |
| 4. | Study I<br>4.1<br>4.2 | Endpoints and Covariates 6 Study Endpoints 6 4.1.1 Primary Endpoint 6 4.1.2 Secondary Endpoints 6 4.1.3 Safety Endpoints 6 Planned Covariates 6 |
| 5. | Hypoth | neses |
| 6. | Definiti<br>6.1<br>6.2<br>6.3<br>6.4<br>6.5 | ions 7 Study Dates 7 Study Points of Reference 8 Baseline and Demographics 8 Efficacy Endpoints 9 Safety Endpoints 9 |
| 7. | Analys<br>7.1<br>7.2<br>7.3<br>7.4<br>7.5 | is Subsets 10 Full Analysis Set 10 Safety Analysis Set 10 Efficacy Analysis Set 10 Per Protocol Set 11 Subgroup Analyses 11 |
| 8. | Interim | Analysis and Early Stopping Guidelines11 |
| 9. | Data S<br>9.1<br>9.2<br>9.3<br>9.4<br>9.5<br>9.6 | Creening and Acceptance |






Product: AMG 334

Statistical Analysis Plan: 20140254

| Date | : 07 Jar | nuary 2017 | Page 3 |
|---|---|---|---|
| | 9.7 | Validation of Statistical Analyses | 13 |
| 10. | Statist | Statistical Methods of Analysis | |
| | 10.1 | General Principles | 14 |
| | 10.2 | Subject Accountability | 14 |
| | 10.3 | Important Protocol Deviations | 14 |
| | 10.4 | Demographic and Baseline Characteristics | 15 |
| | 10.5 | Efficacy Analyses | 15 |
| | | 10.5.1 Analyses of Primary Efficacy Endpoint | 16 |
| | | 10.5.2 Analyses of Secondary Efficacy Endpoints | 17 |
| | 10.6 | Safety Analyses | 18 |
| | | 10.6.1 Adverse Events | 18 |
| | | 10.6.2 Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 |
| | | 10.6.3 Laboratory Test Results | 18 |
| | | 10.6.4 Vital Signs | 19 |
| | | 10.6.5 Antibody Formation | 19 |
| | | 10.6.6 Exposure to Concomitant Medication | 19 |
| | 10.7 | Pharmacokinetic Analysis | 19 |
| | 10.8 | Additional Safety Endpoints for Country Specific Supplement Countries | 20 |
| 11. | Chang | es From Protocol-specified Analyses | 20 |
| 12. | Literat | ure Citations / References | 21 |
| 13. | Data N | lot Covered by This Plan | 22 |
| 14. | Appen | dices | 23 |
| | | List of Tables | |
| Tabl | le 1. Su | mmary of Efficacy Endpoints and Analysis Methods | 16 |
| | | List of Appendices | |
| App | endix A. | Post-baseline Study Visits | 24 |
| App | endix B. | Technical Detail and Supplemental Information Regarding Statistical Procedures and Programs | 25 |
| App | endix C. | Reference Values/Toxicity Grades | 28 |
| Ann | endix D | Concomitant Medications | 29 |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017 Page 4

## **Table of Abbreviations**

| Abbreviation or Term | Definition/Explanation |
|----------------------|----------------------------------------------|
| AFT | Accelerated Failure Time Model |
| ANOVA | Analysis of Variance |
| ANCOVA | Analysis of Covariance |
| CI | Confidence Interval |
| CRF | Case Report Form |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| DMC | Data Monitoring Committee |
| DMP | Data Management Plan |
| DRE | Disease Related Event |
| DTP | Data Transfer Plan |
| EAS | Efficacy Analysis Set |
| ECG | Electrocardiograph |
| EOS | End Of Study |
| ETT | Exercise Treadmill Test |
| ETTr | Exercise Treadmill Test post-randomization |
| FAS | Full Analysis Set |
| HR | Heart Rate |
| IP | Investigational Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI | National Cancer Institute |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| TEAE | Treatment Emergent Adverse Event |
| TET | Total Exercise Time |
| ULN | Upper Limit of Normal |
| VHP | Voluntary Harmonization Procedure |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


#### 1. Introduction

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within Protocol Amendments 4 and associated Country Specific Supplement 3 for AMG 334 Study 20140254 dated 28 October 2016 and 14 November 2016, respectively. The scope of this plan includes the primary and final analyses that are planned and will be executed by the Biostatistics department unless otherwise specified.

## 2. Objectives

## 2.1 Primary

To evaluate the effect of AMG 334 compared to placebo on exercise capacity in subjects with stable angina as measured by total exercise time (TET) during an exercise treadmill test (ETT).

## 2.2 Secondary

To evaluate the effect of AMG 334 compared to placebo during an ETT on the time to the onset of:

- Exercise-induced angina
- ST-segment depression

#### 2.3 Safety

To evaluate the safety and tolerability of AMG 334 in a population with stable angina.

#### 3. Study Overview

#### 3.1 Study Design

This is a phase 2a, multicenter, randomized, double-blind, placebo-controlled study in subjects with stable angina. At least 54 subjects will be randomized in a 1:1 ratio to receive either a single dose of AMG 334 140 mg or placebo intravenously prior to completing an ETT. Randomization will be stratified by the TET average of the 2 qualifying screening ETTs (< 7 minutes or  $\geq$  7 minutes). Treatment group will be blinded to the investigator, subjects, and the Amgen study team.

#### 3.2 Sample Size

The primary endpoint is the change from baseline in TET. Assuming between-subject standard deviation for change from baseline in exercise duration of 130 seconds, with a planned study size of at least 27 subjects in each group and a difference in change from baseline in exercise duration of 0 seconds between AMG 334 group and placebo group, there is an 80% probability (power) that the lower bound of the 90% confidence interval





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


(CI) will exceed -90 seconds. A margin larger than -60 seconds between groups was required to accommodate the possibility of more than 60 second (up to 20%) difference allowed in qualifying TETs for individual subjects. Because of this within-subject TET variation, a maximum TET difference of 90 seconds between the AMG 334 group and placebo group was considered reasonable in this study. A margin of -90 seconds was selected, which corresponds to the margin used in previous study testing a comparable hypothesis (Patterson, et.al 2005). Twenty-nine subjects are needed in each group if considering 5% dropout.

When approximately 45 subjects have been enrolled, Amgen may conduct a blinded sample size-estimation and may choose to alter the sample size based on the blinded variance in the pooled treatment groups.

- 4. Study Endpoints and Covariates
- 4.1 Study Endpoints
- 4.1.1 Primary Endpoint
  - · Change from baseline in TET

#### 4.1.2 Secondary Endpoints

- · During the ETT
  - o Time to onset of exercise-induced angina
  - o Time to onset of ≥ 1 mm ST-segment depression

#### 4.1.3 Safety Endpoints

- Adverse events and disease related events
- Changes in vital signs

For Country Specific Supplement countries only:

- Maximum change in ST-segment depression (mm) from baseline
- Maximum heart rate (HR)
- o Maximum change in systolic blood pressure (SBP) from baseline

#### 4.2 Planned Covariates

The stratification factor of baseline TET (< 7 or  $\ge 7$  minutes) will be included as a covariate in the primary analysis of the efficacy endpoints.

Stratification factor will use the values used for randomization unless otherwise noted.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


## 5. Hypotheses

The primary endpoint of the study will be tested for AMG 334 compared to placebo, with type I error 0.1

- Null Hypothesis: In subjects with angina, AMG 334 does significantly decrease
  exercise capacity (by at least 90 seconds), as measured by change from
  baseline in total exercise time, compared to placebo, and that the true treatment
  difference in change from baseline in TET is -90 seconds or more (worse).
- Alternative Hypothesis: In subjects with angina, AMG334 does not decrease
  exercise capacity, as measured by change from baseline in total exercise time,
  compared to placebo, and that the difference in change from baseline in TET if
  any, is less than a 90 second decrease.

#### 6. Definitions

## 6.1 Study Dates

## **Enrollment Date**

Enrollment Date is defined as the randomization date.

#### **Randomization Date**

Randomization Date is defined as the date subject was allocated to a treatment group.

#### First IP Dose Date

First IP Dose Date is the date on which a subject is administered the first dose of IP following randomization. For subjects who are randomized but not dosed with IP, first dose date is missing.

#### Subject-level End of Study (EOS) Date

End of study for each subject is defined as the last date on which the subject last completed a protocol-specified procedure. The date will be recorded on the End of Study CRF page.

#### **Primary Completion Date**

The primary completion date is defined as the date the last subject completes the on study ETT

## **Study Completion Date**

The study completion date is the EOS date of the last subject in the study.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


## 6.2 Study Points of Reference

#### Study Day 1

Study Day 1 is defined as the first IP dose date. For subjects who are randomized but not dosed, Study Day 1 is defined as the date of randomization.

#### Study Day

Study Day is defined as the number of days from Study Day 1.

Before Study Day 1:

Study Day = (Date of Interest – Date of Study Day 1)

On or after Study Day 1:

Study Day = (Date of Interest – Date of Study Day 1) + 1

Therefore the day prior to Study Day 1 is -1.

#### Post-baseline Study Visit

See Appendix A.

#### **Completing Study**

A subject is defined as completing study if the primary reason for ending study is "Completed".

#### Completing Investigational Product (IP)

A subject is defined as completing IP if the reason for ending IP is "Completed".

#### 6.3 Baseline and Demographics

#### **Age at Enrollment**

Subject age at enrollment will be collected in years in the clinical database.

#### **Baseline Values**

Baseline TET is the average of the 2 qualifying screening ETTs.

If subject completes Columbia-Suicide Severity Rating Scale (C-SSRS) form on Study Day 1 then all individual items from Study Day 1 visit will be used as baseline. If subject does not complete C-SSRS form on Study Day 1 then the last completed form prior to Study Day 1 will be used.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


For all other variables, unless otherwise specified, baseline values are defined as the last non-missing value before the first dose of IP, or randomization date for subjects who never received IP. In cases where baseline measurements are taken on the same day as the first IP dose date, it will be assumed that these measurements are taken prior to IP being administered.

#### **BMI**

Subject's BMI will be derived in kg/m<sup>2</sup> in the clinical database.

## 6.4 Efficacy Endpoints

## **Change from baseline in TET**

Change from baseline in TET = TET from on-study ETT post-randomization - baseline TET

#### **Time to Event**

Time to event (onset of angina, ≥ 1 mm ST-segment depression) is defined as the time subject received IP to the time of event onset.

Time to event = event onset time – time received investigational product

If no event occurs, then subject will be censored at the ETT stop time.

#### 6.5 Safety Endpoints

## **Treatment-Emergent Adverse Event**

Events categorized as adverse events (AEs) starting on or after first dose of IP as determined by the flag indicating if the AEs started prior to the first dose on the Events CRF and up to and including 84 days after the end of IP or end of study, whichever comes first.

Serious adverse events (SAEs) are events categorized as AEs that are starting on or after first dose of IP as determined by the flag indicating if the adverse event started prior to the first dose of the Events CRF and up to and including 84 days after the end of investigational product.

## **Treatment-emergent Disease-related Event**

Events categorized as Disease-related Events (DREs) starting on or after first dose of investigational product as determined by the flag indicated if the event started prior to the first dose on the Events CRF and up to and including 84 days after the end of investigational product.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


Serious disease-related events are events are events categorized as DREs that are starting on or after first dose of investigational product as determined by the flag indicating if the event started prior to the first dose on the Events CRF and up to and including 84 days after the end of investigational product

## Maximum Change from Baseline in SBP

The maximum change from baseline in SBP is calculated by the maximum value of (SBP after first dose date— baseline SBP)

## Maximum Change from Baseline in HR

The maximum change from baseline in HR is calculated by the maximum value of (HR after first dose date — baseline HR)

## Maximum Change from Baseline in ST-Segment Depression

The maximum change from baseline in ST-Segment Depression is calculated by the maximum value of (ST-Segment Depression after first dose—baseline ST-Segment Depression).

#### Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a clinician rating of suicidal behavior and ideation. Two versions depending on the type of visits will be used in this study: Screening and Since Last Visit. The C-SSRS consists of a maximum of 20 items to evaluate suicidal behavior and suicidal ideation.

#### 7. Analysis Subsets

## 7.1 Full Analysis Set

The Full Analysis Set (FAS) includes all randomized subjects. Subjects will be analyzed according to their randomized treatment, regardless of the treatment received.

## 7.2 Safety Analysis Set

The Safety Analysis Set (SAS) includes all randomized subjects who received at least one dose of investigational product. For all safety analyses, subjects will be grouped according to the actual treatment received.

## 7.3 Efficacy Analysis Set

The Efficacy Analysis Set (EAS) utilizes the FAS and includes subjects who received IP and completed the exercise treadmill test post-randomization (ETTr). Subjects will be grouped according to their randomized treatment, regardless of the treatment received.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


#### 7.4 Per Protocol Set

The Per Protocol Set (PPS) utilizes the EAS and includes subjects who completed IP on Study Day 1 and do not have important protocol deviations that will potentially impact primary analysis of efficacy endpoints. Subjects who deviate from key eligibility criteria including currently participating in another investigational device or drug study (exclusion criteria 201) and cardiovascular conditions (exclusion criteria 214, 215, 216, 217, 218) will be excluded from the analysis.

## 7.5 Subgroup Analyses

Primary and secondary analyses will be performed according to the following subgroups: baseline TET (< 7 minutes or  $\geq$  7 minutes) randomization strata, age group (<65,  $\geq$ 65) and sex.

#### 8. Interim Analysis and Early Stopping Guidelines

A Data Monitoring Committee (DMC) will review all available safety data periodically. The DMC will have access to subjects' individual treatment assignments. To minimize the potential introduction of bias to the conduct of the study, members of the DMC will not have any direct contact with study center personnel or subjects. The DMC will communicate major safety concerns and recommendations regarding study modification or termination based on the safety parameters to Amgen in accordance with the DMC charter.

Records of all meetings will be maintained by the DMC for the duration of the study.

Records of all meetings will be stored in the Amgen official document management system at the conclusion of the study. Further details are provided in the DMC charter.

No interim analysis is planned for this study except for sample size re-estimation that will be performed on the pooled sample after 45 subjects have been enrolled. Amgen may choose to alter the sample size based on the pooled variance in the overall group.

## 9. Data Screening and Acceptance

## 9.1 General Principles

The objective of the data screening is to assess the quantity, quality, and statistical characteristics of the data relative to the requirements of the planned analyses.

## 9.2 Data Handling and Electronic Transfer of Data

The Amgen Global Study Operations-Data Management (GSO-DM) department will provide all data to be used in the planned analyses. This study will use the RAVE database. The database will be subjected to edit check outlined in the Data





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


Management Plan (DMP). Central laboratory, PK, antibody, biomarkers, adjudicated events and ECG data is outside of RAVE database. All the datasets to be used for planned analyses will be received from GSO-DM department. Additional details will be provided in the DMP and Data Transfer Plan (DTP).

#### 9.3 Handling of Missing and Incomplete Data

Subjects may miss specific data points for a variety of causes. In general, data could be missing due to a subject's early withdrawal from study, a missed visit, or inability to evaluate an endpoint at a particular point in time. Missing assessment at baseline or on-study will not be imputed.

## 9.3.1 Missing and Incomplete Dates

Missing and partially missing dates for the following parameters will be queried. In general, the algorithm for imputing missing dates will use the logic below. Unless otherwise specified, Study Day 1 will be the first dose date or randomization date for subjects who never received IP:

- If the year and month are the same as Study Day 1 but the day part is missing, the day will be set to the 1<sup>st</sup> of the month of Study Day 1.
- If the year is the same as Study Day 1 but the day and month are missing, the
  day and month will be set to the 1<sup>st</sup> of January of Study Day 1.
- If the year and day are the same as Study Day 1 but month is missing, the month will be set to January of Study Day 1.
- If the month and day are the same as Study Day 1 but year is missing, the year will be reset to the year of Study Day 1.
- If any of the resulting dates are prior to reference date, the imputed date will be reset to the reference date.
- If day, month and year are all missing, no imputation will be applied.

Partial/missing AE and concomitant medication start dates will be imputed using the algorithm above, with the Study Day 1 being the first dose date. For subjects who are randomized but not dosed, Study Day 1 is defined as the date of randomization. AEs that occurred before first dose as indicated by "Did event start before first dose of investigational product" is marked 'Y', will not be imputed.

## 9.4 Detection of Bias

This study has been designed to minimize potential bias by allocating treatment groups randomly, assessing endpoints and handling withdrawals without knowledge of the treatment. Other factors that may bias the results of the study include:





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


 important protocol deviations likely to impact the analysis and interpretation of the efficacy endpoints

- · inadvertent breaking of the blind before formal unblinding
- investigational product dosing non-compliance
- · the timing of and reasons for early withdrawal from treatment and from study

The incidence of these factors may be assessed. Important protocol deviations will be listed and/or tabulated in the clinical study report (CSR). If necessary, the incidence of other factors will be tabulated.

Any breaking of the blind for individual subjects prior to formal unblinding of the study will be documented in the CSR.

#### 9.5 Outliers

Histograms will be examined to identify outliers in any of the continuous variables used in the analyses. Unexpected and/or unexplained values in categorical data will be identified by utilizing frequency tables.

Extreme data points will be identified during blinded review of the data before final database lock. These data points will be reviewed and queried per the data management or clinical listing review plans. Extreme values will not be excluded from the analyses.

#### 9.6 Distributional Characteristics

Statistical assumptions for the primary and secondary endpoint analyses will be assessed. Continuous endpoints of change from baseline in TET will be analyzed under normality assumption. If the assumptions for the primary analysis are not met, then suitable transformation methods (eg, log transform) will be applied.

## 9.7 Validation of Statistical Analyses

Programs will be developed and maintained, and output will be verified in accordance with current risk-based quality control procedures.

Tables, figures, and listings will be produced with validated standard macro programs where standard macros can produce the specified outputs.

The production environment for statistical analyses consists of Amgen-supported versions of statistical analysis software; for example, the SAS System version 9.3 or later.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


#### 10. Statistical Methods of Analysis

#### 10.1 General Principles

The primary analysis to evaluate the effect of AMG 334 compared to placebo on exercise capacity in subjects with stable angina as measured by TET during an ETT.

The FAS will be used to tabulate demographic data, baseline disease characteristics, and subject disposition. The EAS will include all FAS subjects who received IP and completed the ETTr and will be used to analyze the primary and secondary endpoints including the change from baseline in TET, time to onset of ≥ 1 mm ST-segment depression, and time to onset of exercise-induced angina. The Safety Analysis Set will be used to analyze safety endpoints.

Summary statistics by each treatment group will be tabulated at each visit. For continuous endpoints, descriptive statistics will be provided including number of subjects, mean, median, standard deviation, standard error, lower and upper quartiles, minimum, and maximum. For categorical endpoints, frequency, and percentage will be given. Missing data will not be imputed.

Baseline value for exercise duration is the average value of the two qualifying measurements in the screening period.

## 10.2 Subject Accountability

The number and percent of subjects who were screened, randomized, received IP, received partial or none, completed study, discontinued study and reasons for discontinuing will be summarized by treatment group.

The number and percent of subjects randomized will be tabulated by study site.

Key study dates for the first subject enrolled, last subject enrolled, last subject's end of study, and last subject's ETT will be presented.

Data analysis will occur at the following time points:

The primary analysis will take place after all subjects have completed the on study ETT.

The final analysis will take place after all subjects have completed the study and after the final database lock.

#### 10.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined by the study team before the first subject's visit and updated during the IPD reviews throughout the study prior to database lock. These definitions of IPD categories, sub-category codes, and





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


descriptions will be used during the course of the study. Eligibility deviations are defined in the protocol.

## 10.4 Demographic and Baseline Characteristics

Demographic (ie, age, age group (based on median cut point), geriatric age group [< 65, ≥ 65 and ≥75], sex, race, ethnicity) and baseline disease characteristics will be summarized by treatment group and overall using descriptive statistics.

If multiple races have been reported for a subject, the subject will be categorized as multiple race.

The following baseline characteristics will also be summarized:

- Weight (kg)
- Height (cm)
- Body Mass Index (BMI, kg/m2)
- Systolic BP (mmHg)
- Diastolic BP (mmHg)
- Heart Rate (beats/min)
- Baseline TET (seconds)
- Concomitant medications of interest (beta blockers, nitrates, calcium channel blockers, ranolazine, ACE inhibitors and angiotensin receptor blockers)

## 10.5 Efficacy Analyses

Detailed primary, secondary and sensitivity analysis methods are summarized in the table below.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


Table 1. Summary of Efficacy Endpoints and Analysis Methods

| Endpoint | Primary and Secondary<br>Analysis Methods (EAS) | Sensitivity Analysis Methods |
|---|---|---|
| Primary Endpoint | | |
| Change from baseline in TET (seconds) | Primary analysis: Two-Way ANOVA model with terms of treatment group and randomization strata (< 7 or ≥ 7 minutes) | Analysis of covariance (ANCOVA) model with terms of treatment group and baseline TET as a continuous measure Repeat primary analysis using the Per Protocol Analysis Set Repeat primary analysis by subgroups, including baseline TET randomization strata, age group and sex (if sample size permits.) |
| Secondary Endpoints | | |
| Time to onset of exercise-induced angina* (seconds) Time to onset of ≥ 1 mm ST-segment depression (seconds) | Primary analysis: K-M log-rank test stratified by Baseline TET strata (< 7 or ≥ 7 minute) Secondary analysis: Cox proportional hazard model including treatment group and baseline TET as a continuous measure | Repeat primary and secondary analyses using the Per Protocol Analysis Set Repeat primary and secondary analyses by subgroups including baseline TET randomization strata, age group and sex (if sample size permits) |
| | Serial See Model | |

<sup>\*</sup>includes angina-related symptoms

## 10.5.1 Analyses of Primary Efficacy Endpoint

The analysis for the primary endpoint, evaluating change from baseline in TET, will be performed using the EAS. The primary hypothesis is that AMG 334 does not substantially decrease exercise capacity, as measured by change from baseline in exercise duration, compared to placebo (ie, the true treatment difference in change from baseline in exercise duration is -90 seconds or more).

In the primary analysis, the primary endpoint will be analyzed using an ANOVA model with terms for treatment group and baseline TET (< 7 or  $\geq$  7 minutes) randomization strata. Adjusted group means for each treatment group, standard error, 90% CI, difference of group means compared to placebo and associated 90% CIs will be tabulated. If the lower bound of the 90% CI of the difference is more than -90 seconds, then the hypothesis that AMG 334 does not substantially decrease exercise duration will be supported.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


Statistical assumptions for the primary endpoint method of analysis will be assessed. If the assumptions for the primary analysis are not met, then nonparametric methods or suitable transformation will be utilized.

Sensitivity analyses described below will be performed for the primary endpoint using the EAS:

- An analysis of covariance (ANCOVA) model including treatment group and baseline TET as a continuous measure
- The primary analysis will be repeated using the PPS

To assess if the treatment effect varies across subgroups of interest, the primary analysis of the primary endpoint will be repeated and will include an interaction term (treatment group\* subgroup) in the ANOVA model. If a treatment group\*subgroup interaction is observed at a significance level of 0.10, then the primary analysis may be repeated for each level of the subgroup. In addition, reasons for stopping the ETTr will be summarized by treatment group using the EAS.

## 10.5.2 Analyses of Secondary Efficacy Endpoints

The secondary endpoints are time to onset of exercise-induced angina and time to onset of  $\geq 1$  mm ST-segment depression.

For time-to-event endpoints, only the first occurrence will be considered. If no event is observed during ETTr, then this subject will be considered as censored at the end of ETTr.

Kaplan-Meier estimates of the event-free time to ST-segment depression and exercise induced angina will be computed and graphically displayed using the EAS. For each endpoint, a stratified (< 7 or ≥ 7 minute randomization strata) log-rank test statistic will be calculated to compare the two treatment groups at a significance level of 0.10.

As a secondary analysis, the hazard ratio and its 90% CI for AMG 334 vs placebo will be estimated using a stratified (< 7 or ≥ 7 minute randomization strata) Cox proportional hazards regression model. The proportional hazards assumption will be assessed by visual inspection for parallel lines over time in the plot of log-negative-log of the survival function vs. log (time) (Hosmer and Lemeshow, 1999). If there is strong evidence of non-proportional hazards for the treatment group, then a piece-wise Cox model (Collett, 2003) or an accelerated failure time (AFT) model will be considered. Regardless of non-proportionality, the main analysis of the primary endpoint will be in terms of the Cox model.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


Summary statistics (mean, median, Q1, Q3, and 90% CI) of time to event will be provided by treatment group. The number and percentage of subjects with an observed event will also be provided.

Sensitivity analyses described below will be performed for the secondary endpoints:

 Repeat the secondary analysis (Cox proportional hazards regression) using baseline TET as a continuous measure

Repeat the primary and secondary analysis using PPS

#### 10.6 Safety Analyses

#### 10.6.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) version 18.0 or later will be used to code all events categorized as AEs and Disease-related Events (DREs) to a system organ class and a preferred term.

Subject incidence of AEs will be summarized for all treatment-emergent AEs, serious AEs, AEs leading to withdrawal of IP and fatal AEs. Subject incidence of all treatment-emergent AEs, serious AEs, AEs leading to withdrawal of IP and fatal AEs, will be tabulated by system organ class and preferred term in descending order of frequency. Subgroups group analyses (if there is a medical rationale) will be presented by system organ class and preferred term in descending order of frequency. All races (if appropriate) with less than 5% of the total enrolled subjects will be pooled together for summary purposes.

Subject-level data may be provided instead of tables if the subject incidence is low.

Subject incidence of DREs will be summarized for all treatment-emergent DREs and fatal DREs.

## 10.6.2 Columbia-Suicide Severity Rating Scale (C-SSRS)

No statistical testing will be performed on C-SSRS. The number and percentage of subjects reporting any suicidal ideation and any suicidal behavior will be summarized descriptively by treatment group. Shift table of C-SSRS maximum severity of suicidal ideation/behavior compared to baseline will be provided by treatment group.

#### 10.6.3 Laboratory Test Results

Shifts tables of the laboratory toxicity for selected lab analytes (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, creatinine) based on Common Terminology Criteria for Adverse Events (CTCAE) grade (version 4) relative to baseline will be tabulated by treatment group for entire study





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


period. In the cases when CTCAE grading scales include numeric ranges in combination with clinical assessment (eg, Potassium [Hypokalemia]), laboratory test results may be summarized based on standard normal ranges or by CTCAE grade utilizing investigator's input.

Summary of change from baseline for absolute neutrophil count (ANC), alanine transaminase (ALT), aspartate aminotransferase (AST) and creatinine will also be provided.

Additional liver test summary table will provide the number and percentage of subjects by treatment group for the following categories:

- AST and ALT ( > 3x ULN; > 5x ULN; > 10x ULN; > 20x ULN respectively)
- AST or ALT ( > 3x ULN; > 5x ULN; > 10x ULN; > 20x ULN respectively)
- Total Bilirubin (> 1x ULN; >1.5x ULN; >2x ULN respectively)
- ALP (>1.5 ULN)
- ALT or AST > 3x ULN and Total Bili ≥ 2x ULN and ALP < 2x ULN

#### 10.6.4 Vital Signs

Descriptive summaries of blood pressures and HR will be provided at baseline and at each study visit. In addition, blood pressures and HR collected during ETTr will be summarized at specific time points (baseline, peak and last measurement). Descriptive summaries will be provided for the maximum change from baseline in SBP and HR on day 1 post dose during ETTr for Country Specific Supplement countries.

#### 10.6.5 Antibody Formation

The incidence and percentage of subjects who develop anti-AMG334 antibodies (binding and if positive, neutralizing) at any time will be tabulated by treatment group.

#### 10.6.6 Exposure to Concomitant Medication

Number and proportion of subjects receiving therapies of interest will be summarized by category for each treatment group as coded by the World Health Organization Drug (WHODRUG) dictionary. See Appendix D for a list of selected medications and their groupings.

#### 10.7 Pharmacokinetic Analysis

All PK-related tables, figures, listings and other deliverables will be generated by PKDM. Serum AMG 334 concentrations will be summarized using descriptive statistics.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


# 10.8 Additional Safety Endpoints for Country Specific Supplement Countries

This section is for countries that were originally aligned with EU VHP (European Union Voluntary Harmonization Procedure) requirements. These countries are listed in the Country Specific supplements of the protocol (ie, Czech Republic, Latvia, Romania, Bulgaria and Poland).

After the end of ETT, all subjects will be followed at the site for at least 4 hours. At the end of the 4-hour follow-up period, the following procedures will be performed:

- 12-lead rest ECG in a sitting position
- Blood pressure measurement in a sitting position
- Blood sampling for measurement of cardiac biomarker (troponin I)

Additional visits for anti-AMG334 antibody (Day1 Pre-dose, week 4, and week 12) and C-SSRS (visit 2, visit 3, visit 4, and week 2) will be collected for countries listed in Country Specific Supplement.

These additional data will be included in the analysis.

## 11. Changes From Protocol-specified Analyses

There are no changes to the protocol-specified analyses.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


#### 12. Literature Citations / References

- O'Brien, R. G. (1981), "A Simple Test for Variance Effects in Experimental Designs," Psychological Bulletin, 89, 570–574.
- Freund, R. J., Littell, R. C., and Spector, P. C. (1986), SAS System for Linear Models, 1986 Edition, Cary, NC: SAS Institute Inc
- Gibbons, J. D. and Chakraborti, S. (1992), Nonparametric Statistical Inference, Third Edition, New York: Marcel Dekker.
- Allison PA. Survival Analysis Using SAS A Practical Guide. SAS Institute Inc.; 1995.
- Brookmeyer R, Crowley J. A confidence interval for the median survival time.
   Biometrics 1982; 38; 29-41.
- Carroll KJ. Analysis of progression-free survival in oncology trials: some common statistical issues. Pharmaceutical Statistics 2007; 6; 99-113.
- Hosmer & Lemeshow Applied Survival Analysis 2nd edition; 2008Collett, David. Modelling Survival Data in Medical Research Gold M, Washington Panel on Cost Effectiveness in Health and Medicine, Med Care, 1996;34(12 Suppl):DS197-9. Boca Raton, FL: Chapman & Hall/CRC, 2003.
- Patterson D, Kloner R, Effron M, et al. The effect of tadalafil on the time to exercise-induced myocardial ischaemia in subjects with coronary artery disease. Br J Clin Pharmacol. 2005, 60: 459-468.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


## 13. Data Not Covered by This Plan

There are no plans to specifically analyze or summarize the following data points.

- Pk
- Data for biomarker development





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017


14. Appendices





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


#### Appendix A. Post-baseline Study Visits

Since the actual visit for a subject may not exactly coincide with their targeted visit date, the actual visit date is mapped to the study visit as following. The study day window will be utilized to define study visit for labs, antibody, vital signs and physical measurements collected at office visits.

| Study Visit | Target Day | Study Day |
|-------------|------------|---------------------------------------------------|
| Week 4 | 29 | 16-43 |
| Week 8 | 57 | 44-71 |
| Week 12 | 85 | 72 to Min (EOS Date, last IP dose date + 84 days) |

#### Note:

- 1. If more than one visit (including unscheduled visits, ie, CPEVENT = 'UNSCHED') fall within the same defined window, scheduled visit will be used regardless of the distance from the target day. Unscheduled visit will only be used when there is no scheduled visit in the defined window. The closest visit to the target day among the same type of visit (scheduled vs. unscheduled) will be considered for analysis. If two assessment dates are equidistant from the target date, the latter visit will be considered for analysis.
- 2. For Country Specific Supplement countries, CSSRS and ECG data are collected at week 2 (target day 14), corresponding to study day 1-28.





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


# Appendix B. Technical Detail and Supplemental Information Regarding Statistical Procedures and Programs

## **Code Fragments**

#### **Section 10.5.1**





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017 Page 26





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017








Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


## Appendix C. Reference Values/Toxicity Grades

Adverse event severity and laboratory parameters are graded based on National Cancer Institute (NCI) Common Toxicity Criteria version 4 or higher, which is available at the following: http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-

14\_QuickReference\_5x7.pdf





Clinical Study Report: 20140254 Primary Analysis

Page 30 Date: 13 April 2017

Product: AMG 334

Statistical Analysis Plan: 20140254 Date: 07 January 2017 Page 29

## Appendix D. Concomitant Medications

| Beta-blockers Beta-blockers BETA BLOCKING AGENTS ADAPROLOL ANTIARRHYTHMIC AGENTS BETA BLOCKING AGENTS BUFETOLOL BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL MOPROLOL MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL ALPRENOLOL ALPRENOLOL ALPRENOLOL BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED 102298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL BOPINDOLOL BUCINDOLOL BUCINDOLOL BUCINDOLOL BUCINDOLOL BUGINDOLOL BUFURALOL BUNITROLOL HYDROCHLORIDE BUNITROLOL BUNITROLOL BUNITROLOL BUNITROLOL BUNITROLOL BUNITROLOL HYDROCHLORIDE | Appendix D. Concomitant Medications | |
|---|---|---|
| ADAPROLOL ANTIARRHYTHMIC AGENTS BETA BLOCKING AGENTS BUFETOLOL BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL | Group | Medications |
| ANTIARRHYTHMIC AGENTS BETA BLOCKING AGENTS BUFETOLOL BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL | Beta-blockers | BETA BLOCKING AGENTS |
| BETA BLOCKING AGENTS BUFETOLOL BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL | | ADAPROLOL |
| BUFETOLOL BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL ALPRENOLOL ALPRENOLOL ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL BUCINDOLOL HYDROCHLORIDE BUCINDOLOL BUCINDOLOL BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL | | ANTIARRHYTHMIC AGENTS |
| BUFETOLOL HYDROCHLORIDE DILEVALOL DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | BETA BLOCKING AGENTS |
| DILEVALOL DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | BUFETOLOL |
| DILEVALOL HYDROCHLORIDE ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL NIFENALOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN BOPINDOLOL BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | BUFETOLOL HYDROCHLORIDE |
| ISAMOLTAN MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | DILEVALOL |
| MABUTEROL MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL | | DILEVALOL HYDROCHLORIDE |
| MABUTEROL HYDROCHLORIDE MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | ISAMOLTAN |
| MOPROLOL MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | MABUTEROL |
| MOPROLOL HYDROCHLORIDE NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | MABUTEROL HYDROCHLORIDE |
| NADOXOLOL NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | MOPROLOL |
| NADOXOLOL HYDROCHLORIDE NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL | | MOPROLOL HYDROCHLORIDE |
| NIFENALOL NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL | | NADOXOLOL |
| NIFENALOL HYDROCHLORIDE OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL | | NADOXOLOL HYDROCHLORIDE |
| OBERADILOL ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUNITROLOL | | NIFENALOL |
| ALPRENOLOL ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | NIFENALOL HYDROCHLORIDE |
| ALPRENOLOL BENZOATE ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL | | OBERADILOL |
| ALPRENOLOL HYDROCHLORIDE BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL BUFURALOL BUFURALOL | | ALPRENOLOL |
| BETA BLOCKING AGENTS, NON-SELECTIVE BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL | | ALPRENOLOL BENZOATE |
| BETAMED /02298401/ BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL | | ALPRENOLOL HYDROCHLORIDE |
| BLOCOTIN /00716001/ BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL HYDROCHLORIDE | | BETA BLOCKING AGENTS, NON-SELECTIVE |
| BOPINDOLOL BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL HYDROCHLORIDE | | BETAMED /02298401/ |
| BOPINDOLOL FUMARATE BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUFURALOL HYDROCHLORIDE BUNITROLOL | | BLOCOTIN /00716001/ |
| BOPINDOLOL MALONATE BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUNITROLOL | | BOPINDOLOL |
| BUCINDOLOL BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUNITROLOL | | BOPINDOLOL FUMARATE |
| BUCINDOLOL HYDROCHLORIDE BUFURALOL BUFURALOL HYDROCHLORIDE BUNITROLOL | | BOPINDOLOL MALONATE |
| BUFURALOL BUFURALOL HYDROCHLORIDE BUNITROLOL | | BUCINDOLOL |
| BUFURALOL HYDROCHLORIDE BUNITROLOL | | BUCINDOLOL HYDROCHLORIDE |
| BUNITROLOL | | BUFURALOL |
| | | BUFURALOL HYDROCHLORIDE |
| BUNITROLOL HYDROCHLORIDE | | BUNITROLOL |
| | | BUNITROLOL HYDROCHLORIDE |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**BUPRANOLOL** 

**BUPRANOLOL HYDROCHLORIDE** 

CARAZOLOL CARTEOLOL

CARTEOLOL HYDROCHLORIDE

**CLORANOLOL** 

**CLORANOLOL HYDROCHLORIDE** 

CLOTAS PLUS EXAPROLOL

**EXAPROLOL HYDROCHLORIDE** 

**INDENOLOL** 

INDENOLOL HYDROCHLORIDE

**MEPINDOLOL** 

MEPINDOLOL SULFATE

**METIPRANOLOL** 

METIPRANOLOL HYDROCHLORIDE

NADOLOL NIPRADOLOL

**OXPRENOLOL** 

OXPRENOLOL HYDROCHLORIDE

**PENBUTOLOL** 

PENBUTOLOL SULFATE

PINDOLOL PRONETALOL

PRONETALOL HYDROCHLORIDE

**PROPRANOLOL** 

PROPRANOLOL HYDROCHLORIDE PROPRANOLOL PHENOBARBITAL

SOLOPOSE BETA SOTACOR/ASA

SOTALOL

SOTALOL HYDROCHLORIDE

TENSYN PLUS TERTATOLOL

TERTATOLOL HYDROCHLORIDE

**TILISOLOL** 





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


TILISOLOL HYDROCHLORIDE

TIMOLOL

TIMOLOL HEMIHYDRATE

TIMOLOL MALEATE

TIMOLOL MALEATE, R-ENANTIOMER
TIMOLOL MALEATE, S-ENANTIOMER
ZEPRO /02777801/

**ACEBUTOLOL** 

ACEBUTOLOL HYDROCHLORIDE

**ATENOLOL** 

ATENOLOL HYDROCHLORIDE

BELOC /01739801/

BETA BLOCKING AGENTS, SELECTIVE

**BETAXOLOL** 

BETAXOLOL HYDROCHLORIDE

**BEVANTOLOL** 

BEVANTOLOL HYDROCHLORIDE

**BISOBLOCK PLUS** 

**BISOPROLOL** 

**BISOPROLOL FUMARATE** 

**BUCUMOLOL** 

BUCUMOLOL HYDROCHLORIDE

BUTIDRINE

**CELIPROLOL** 

CELIPROLOL HYDROCHLORIDE

**DEXNEBIVOLOL** 

DIACETOLOL

DIACETOLOL HYDROCHLORIDE

**EPANOLOL** 

**ERAMID** 

**ESATENOLOL** 

**ESMOLOL** 

ESMOLOL HYDROCHLORIDE

LANDIOLOL

LANDIOLOL HYDROCHLORIDE

LEVONEBIVOLOL





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**METOPROLOL** 

METOPROLOL SUCCINATE
METOPROLOL TARTRATE
METOPROLOL W/MORPHINE

METPURE ST

**NEBIVOLOL** 

NEBIVOLOL HYDROCHLORIDE

**PAFENOLOL** 

**PRACTOLOL** 

SELOKEN ZOC/ASA

TALINOLOL

**TOLAMOLOL** 

TOLAMOLOL HYDROCHLORIDE

ZOLAT /03453901/

ALPHA AND BETA BLOCKING AGENTS

AMINO ACIDS NOS W/CAFFEINE/CARVEDILOL/CHOLINE

**AMOSULALOL** 

AMOSULALOL HYDROCHLORIDE

**AROTINOLOL** 

AROTINOLOL HYDROCHLORIDE

CARVEDILOL

CARVEDILOL HYDROCHLORIDE

CARVEDILOL PHOSPHATE HEMIHYDRATE

LABETALOL

LABETALOL HYDROCHLORIDE

**MEDROXALOL** 

MEDROXALOL HYDROCHLORIDE

PROXODOLOL

BETA BLOCKING AGENTS AND THIAZIDES

BETA BLOCKING AGENTS, NON-SELECTIVE, AND THIA

**BETACENTYL** 

CORGARETIC

**CORINDOCOMB** 





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**DOCIDRAZIN** 

HIPERDON /00991401/

INDERETIC

**INDERIDE** 

**PRESTYL** 

**SOTAZIDE** 

**TIMOLIDE** 

**TORRAT** 

**TRASIDREX** 

TRI-TORRAT

VISKAZIDE

ATENOLOL W/HYDROCHLOROTHIAZIDE

ATPURE-D

**BELOC-ZOC COMP** 

BETA BLOCKING AGENTS, SELECTIVE, AND THIAZIDE

BISELECT /01166101/

BISOPROLOL W/HYDROCHLOROTHIAZIDE /06833601/

CO-BETALOC

**NEATENOL DIU** 

**NEATENOL DIUVAS** 

**NEBICARD-H** 

**RANEZIDE** 

SECADREX

SECTRAZIDE /00774201/

SELOKEN COMP.

**TRELOC** 

ALPHA AND BETA BLOCKING AGENTS AND THIAZIDES

CO-DILATREND

NORMOZIDE /00897401/

BETA BLOCKING AGENTS AND OTHER DIURETICS

BETA BLOCKING AGENTS, NON-SELECTIVE/90118901/

**BETARELIX** 

HIPERDON /00991401/





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**LASIPRESSIN** 

**SANDORETIC** 

**SPIROPROP** 

**TRASITENSIN** 

**TREPRESS** 

VISKALDIX

BETA BLOCKING AGENTS, SELECTIVE, AND OTHER DI

INDAPAMIDE W/NEBIVOLOL HYDROCHLORIDE

**LOPRESORETIC** 

NOR-PA

SALI-PRENT

**SELECTURON** 

**TEKLO** 

**TENORETIC** 

TRI-NORMIN

VINICOR D

ALPHA AND BETA BLOCKING AGENTS AND OTHER DIUR

CARVEDILOL + CLORTALIDONA

**TRANDIUR** 

BETA BLOCKING AGENTS, THIAZIDES AND OTHER DIU

BETA BLOCKING AGENTS, NON-SELECTIVE, THIAZIDE

CARDIOTENSIN /01682501/

**DOCITEREN** 

DOCITON 80 DYTIDE H

MODUCREN

BETA BLOCKING AGENTS, SELECTIVE, THIAZIDES AN

**KALTEN** 

KERLIDEX

BETA BLOCKING AGENTS AND VASODILATORS

BETA BLOCKING AGENTS, NON-SELECTIVE, AND VASO

**BETA-INTENSAIN** 

**NITRISKEN** 

NITRO-OBSIDAN





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


OXYCARDIN /00391901/

**PRIZIDILOL** 

PRIZIDILOL HYDROCHLORIDE

PRIZIDILOL HYDROCHLORIDE ANHYDROUS

BETA BLOCKING AGENTS, SELECTIVE, AND VASODILA

MET XL R

METOPROLOL W/RAMIPRIL

NEBICARD V

STARPRESS R

BETA BLOCKING AGENTS AND OTHER ANTIHYPERTENSI

BETA BLOCKING AGENTS, NON-SELECTIVE/90119501/

**BETADIPRESAN** 

**INDUCOR** 

INDUCOR D

OBSILAZIN

REDUPRESS /03518901/

TRASIPRESSOL

TRIMECRYTON

AMLODIPINE W/METOPROLOL

AMLODIPINE W/NEBIVOLOL

AMLONG-A

ARBITEL MT

ATPURE-SA

**BELNIF** 

BETA BLOCKING AGENTS, SELECTIVE, AND OTHER AN

BETAFIT AM

**BETAONE AM** 

**CARDIF BETA** 

CARDIORETIC A

CARVEDIPINA D

CILNIDIPINE W/METOPROLOL SUCCINATE

CILNIPAR M

**CONCOR AM** 




Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**CONCORAM** 

FELODIPINE W/METOPROLOL

**FIXOCARD** 

LOTENSYL AT

MET XL AM

METONCE AM

METOPROLOL W/TELMISARTAN

**MODILOC** 

NEBI AM

**NEBICARD-SM** 

NIF-TEN

**NITRENOL** 

**NUSAR-ATN** 

OLSAR M

**RASOTAN BETA** 

**TELISTA MT** 

**TONORMA** 

**TREDALAT** 

**ADAPROLOL** 

ALCON BETAXOLOL

**AZARGA** 

BAMOSIRAN

BEFUNOLOL

BEFUNOLOL HYDROCHLORIDE

BETA BLOCKING AGENTS

BETALOL /03186001/

**BETAXOLOL** 

BETAXOLOL HCL W/PILOCARPINE HCL

BETAXOLOL HYDROCHLORIDE

BETAXOLOL W/PILOCARPINE

BLOCANOL /01100601/

BRIMONIDINE TARTRATE W/TIMOLOL

BRIMONIDINE W/TIMOLOL





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


CARPILO

CARTEOL /00853401/

CARTEOLOL

CARTEOLOL HYDROCHLORIDE

CARTEOPIL COMBIGAN COSOPT

DORZOLAMIDE W/TIMOLOL

DORZOPT /06421101/

DUOTRAV ELAZOP GANFORT

GLAUTIMOL /06108601/

KRITANTEK OFTENO KRYTANTEK OFTENO

LEVOBUNOLOL

LEVOBUNOLOL HYDROCHLORIDE

METIPRANOLOL

METIPRANOLOL HYDROCHLORIDE

**MOPROLOL** 

MOPROLOL HYDROCHLORIDE

NIPRADOLOL

NORMOGLAUCON /01482401/

PILOBLOQ
PILOFLAX
PINDOLOL
PROXODOLOL
PROXOPHELIN

**RIPIX** 

TAFLUPROST W/TIMOLOL MALEATE

TIMED
TIMOLO
TIMOLOL





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

| | TIMOLOL HEMIHYDRATE |
|----------|--------------------------------------------------|
| | TIMOLOL MALEATE |
| | TIMOLOL MALEATE, R-ENANTIOMER |
| | TIMOLOL MALEATE, S-ENANTIOMER |
| | TIMPILO |
| | VISTAGAN /00844001/ |
| | XALACAR-T |
| | XALACOM |
| | ADOCOR /01266201/ |
| Nitrates | ANGIOCARDYL N |
| | ANGOR |
| | ASPITRATE G |
| | BIDIL |
| | CAFINITRINA /00702101/ |
| | CAFINITRINA /07893501/ |
| | CAFINITRINA RETARD |
| | CARDIACAP A |
| | CARDIOSEDANTOL |
| | CEFAVORA COR /08009401/ |
| | CONVALLARIA MAJALIS W/GLYCERYL<br>TRINITRATE/LEV |
| | CORANGIL |
| | DILCORAN /00119101/ |
| | ERITRITYL TETRANITRATE |
| | ERYTHROMIN /01950501/ |
| | EUCARDIN |
| | GLYCERYL TRINITRATE |
| | GLYCERYL TRINITRATE, COMBINATIONS |
| | GOVIL |
| | IMAZIN XL |
| | ISO-NITROLINGUAL |
| | ISOSORBIDE DINITRATE |
| | ISOSORBIDE DINITRATE W/SODIUM CHLORIDE |
| | ISOSORBIDE DINITRATE, COMBINATIONS |
| | ISOSORBIDE MONONITRATE |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**KORDILAT** 

MANNITOL HEXANITRATE

METHYLPROPYLPROPANEDIOL DINITRATE

**MYANGIN** 

 MYOCARDON
 /00091601/

 MYOCARDON
 /02403401/

 MYOCARDON
 /03439401/

MYOCORIL

NATIROSE /01832701/

NEO-AKTAL

NITRANGIN COMPOSITUM

NITRAPAMIL
NITRIC OXIDE

NITRO-CRATAEGUTT

**NITRODURAT** 

**NITROGLIN** 

NITROGLYCERIN COMP.

NITROPENT COMP.

**NITROTHESAL** 

NITROUS ETHER SPIRIT

NUNZANGIL

**ORGANIC NITRATES** 

PENTAERITHRITYL TETRANITRATE

PENTANEURAL

**PENTOXYLON** 

**PENTRINITROL** 

**PENTRIUM** 

PROPATYLNITRATE

SEDA-ILDAMEN

SORBANGIL COMP.

**SPASMOCOR** 

**STENODILATE** 

**STENOPTIN** 

**TENITRAMINE** 

THEOPENTRIT

THEOPENTRIT PAPAV





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

| | TRINITRINE CAFFEINE |
|-----------------|------------------------------------|
| | TROLNITRATE |
| | TROLNITRATE PHOSPHATE |
| | VISANOCOR |
| | VISANOCOR N |
| Calcium channel | VERAPAMIL |
| blockers | VERAPAMIL HYDROCHLORIDE |
| bioditoro | ISOPTIN S |
| | TALUVIAN /00149301/ |
| | LIDOFLAZINE |
| | PERHEXILINE |
| | PERHEXILINE MALEATE |
| | GRADULON |
| | FENDILINE |
| | FENDILINE HYDROCHLORIDE |
| | NIFEDIPINE |
| | DILTIAZEM |
| | DILTIAZEM HYDROCHLORIDE |
| | DILTIAZEM MALATE |
| | DIGO-SENSIT |
| | STENOPTIN |
| | CORDICHIN |
| | ELTHON /00603601/ |
| | NICARDIPINE |
| | NICARDIPINE HYDROCHLORIDE |
| | GALLOPAMIL |
| | GALLOPAMIL HYDROCHLORIDE |
| | FELODIPINE |
| | ISRADIPINE |
| | TIAPAMIL |
| | SALI-ADALAT |
| | BEPRIDIL |
| | BEPRIDIL HYDROCHLORIDE MONOHYDRATE |
| | NITRENDIPINE |
| | TREDALAT |
| | NISOLDIPINE |
| | NIF-TEN |
| | BELNIF |
| | NIMODIPINE |
| | VERATIDE |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**OXODIPINE** 

**AMLODIPINE** 

AMLODIPINE BESILATE
AMLODIPINE MALEATE
AMLODIPINE MESILATE
AMLODIPINE CAMSILATE
AMLODIPINE OROTATE
S AMLODIPINE NICOTINATE

NILVADIPINE

AMLODIPINE ADIPATE

MANIDIPINE

MANIDIPINE HYDROCHLORIDE

LACIDIPINE BENIDIPINE

BENIDIPINE HYDROCHLORIDE

MODILOC EFONIDIPINE

EFONIDIPINE HYDROCHLORIDE

SALOPTASIN BARNIDIPINE

BARNIDIPINE HYDROCHLORIDE

UDRAMIL MIBEFRADIL

MIBEFRADIL HYDROCHLORIDE

LEXXEL

TECZEM /01366001/

LERCANIDIPINE

LERCANIDIPINE HYDROCHLORIDE

CILNIDIPINE VERACAPT UNIMAX

ADIZEM-XL PLUS

ANIPAMIL TILDIAZIDE

OCADRIK /01507301/

AZELNIDIPINE

**ENEAS** 

NIMOREAGIN /01616501/

AMLODIPINE W/BENAZEPRIL

AMLODIPINE BESYLATE W/BENAZEPRIL

AMLODIPINE W/VALSARTAN





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


AMLODIPINE W/HYDROCHLOROTHIAZIDE

AMLONG-A CADUET ARANIDIPINE

SINERGEN

HYDROCHLOROTHIAZIDE W/VERAPAMIL

LOTAR /02225901/

AMLOPRES L RIODIPINE DIOVAN AMLO MET XL AM TONORMA FIXOCARD

LOTRIX /03460001/

NIMOSOMAZINA

REDUPRESS /03518901/

NAPRIX A
ASOMEX-D
CARDIF BETA
LOTENSYL AT
ATPURE-SA
NEBICARD-SM
ACEDIP
CLEVIDIPINE
ANTROLIN
CARDIORETIC A
NITRENOL
ETIPRESS-D

MAXIDIPIN DIU NIFEDIP D CARVEDIPINA D

INDUCOR INDUCOR D BETAONE AM

AZOR /06230801/

AMLOZAAR-H TWYNSTA TELSAR-A DIOVAN TRIPLE OROSPREVENT COVERAM





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


NEMOCEBRAL PLUS

LEVAMLODIPINE

LEVAMLODIPINE BESILATE
LEVAMLODIPINE MALATE
LEVAMLODIPINE MALEATE
FELODIPINE W/METOPROLOL
NIFEDIPINE W/TELMISARTAN

PONTUC DIRONORM COZAAR XQ

BENITEC A /06541301/

OLMESAFE AM CONCOR AM CANDESAR A

AMLODIPINE W/ATORVASTATIN

TRIBENZOR ATACAND DUO

AMLODIPINE MALEATE W/BENAZEPRIL

HYDROCHLORIDE RASILEZ AMLO AMTAS PRP FLORDIPINE NIGULDIPINE NORVERAPAMIL AZIDOPINE

AMLODIPINE W/BENAZEPRIL HYDROCHLORIDE

VIVACE /06864501/

FENSARTAN UNIMAX

AMTURNIDE

**IGANIDIPINE** 

**AVOTIN** 

AZELNIDIPINE W/OLMESARTAN MEDOXOMIL

AMLODIPINE BESILATE W/ATORVASTATIN CALCIUM

TR

MOXOVAS A OLMAT AMH

TEKAMLO /07156301/

AMI ODIPINE

W/HYDROCHLOROTHIAZIDE/VALSARTAN

NATRILAM BETAFIT AM CILACAR T





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


MODLIP AM

**NEBI AM** 

**DILVAS AM** 

R PRIL AM

AMLODAC D

**TELMICHEK AH** 

**RASITRIO** 

**DUPLECOR** 

PERINDOPRIL ARG/AMLODIPINE FISHER

**CONCORAM** 

**AMLATOR** 

TAH

**ENALAPRIL W/NITRENDIPINE** 

**APROVASC** 

COROVAL B

ZANERIL

ENALAPRIL W/LERCANIDIPINE

AMLODIPINE W/OLMESARTAN

**ANOBLISS** 

ASOMEX TM

RAMI ASOMEX

CILNIPAR M

ASOMEX LTH

METONCE AM

**ROSUCOR PLUS** 

AMLODIPINE W/NEBIVOLOL

AMLODIPINE W/INDAPAMIDE/PERINDOPRIL

LERCANIDIPINE HYDROCHLORIDE W/VALSARTAN

LEVAMLODIPINE BESILATE W/VALSARTAN

AMLODIPINE W/CHLORTALIDONE/LOSARTAN

**POTASSIUM** 

CILNIDIPINE W/OLMESARTAN MEDOXOMIL

AMLODIPINE OROTATE W/VALSARTAN

HYDROCHLOROTHIAZIDE W/LEVAMLODIPINE

**BESILATE** 

AMLODIPINE MESILATE

W/HYDROCHLOROTHIAZIDE/VAL

AMLODIPINE W/CHLORTALIDONE/OLMESARTAN

**MEDOXOM** 

AMLODIPINE W/CHLORTALIDONE/TELMISARTAN

AMLODIPINE BESILATE W/INDAPAMIDE/PE/08715301/

AMLODIPINE BESILATE W/PERINDOPRIL TOSILATE

AMLODIPINE BESILATE W/INDAPAMIDE/PE/08717501/





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

| | <del>_</del> |
|---|---|
| | CILNIDIPINE W/VALSARTAN |
| | AMLODIPINE BESILATE W/AZILSARTAN |
| | ATORVASTATIN CALCIUM W/LEVAMLODIPINE<br>BESILATE |
| | CILNIDIPINE W/METOPROLOL SUCCINATE |
| | AMLODIPINE W/METOPROLOL |
| | AMLODIPINE BESILATE W/CANDESARTAN CILEXETIL/H AMLODIPINE W/LISINOPRIL/ROSUVASTATIN |
| | AMLODIPINE W/ROSUVASTATIN |
| | AMLODIPINE ADIPATE W/VALSARTAN |
| | AMLODIPINE W/CLOPIDOGREL BISULFATE |
| | CHLORTALIDONE W/CILNIDIPINE/TELMISARTAN |
| | AMLODIPINE OROTATE W/OLMESARTAN MEDOXOMIL CALCIUM CHANNEL BLOCKERS |
| | SELECTIVE CALCIUM CHANNEL BLOCKERS WITH MAINL |
| | DIHYDROPYRIDINE DERIVATIVES |
| | SELECTIVE CALCIUM CHANNEL BLOCKERS WITH DIREC |
| | PHENYLALKYLAMINE DERIVATIVES |
| | BENZOTHIAZEPINE DERIVATIVES |
| | NON-SELECTIVE CALCIUM CHANNEL BLOCKERS |
| Ranolazine | Ranolazine |
| ACE inhibitors | CAPTOPRIL |
| 7.0E IIIIIbilois | ENALAPRIL |
| | ENALAPRIL MALEATE |
| | CAPOZIDE |
| | PERINDOPRIL |
| | PERINDOPRIL ERBUMINE |
| | PERINDOPRIL ARGININE |
| | PERINDOPRIL TOSILATE |
| | QUINAPRIL |
| | QUINAPRIL HYDROCHLORIDE |
| | CILAZAPRIL |
| | CILAZAPRIL MONOHYDRATE |
| | RAMIPRIL |
| | LISINOPRIL |
| | LISINOPRIL DIHYDRATE |
| | VASERETIC |
| | SPIRAPRIL |
| | SPIRAPRIL HYDROCHLORIDE |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


BENAZEPRIL

BENAZEPRIL HYDROCHLORIDE

**FOSINOPRIL** 

FOSINOPRIL SODIUM

**ENALAPRILAT** 

ZOFENOPRIL

ZOFENOPRIL CALCIUM

ALACEPRIL

**DELAPRIL** 

DELAPRIL HYDROCHLORIDE

**GEZOR** 

**TRANDOLAPRIL** 

**CIBADREX** 

SALUTEC

ARELIX ACE

DYNORM PLUS

QUINAPRILAT

QUINAPRILAT HYDRATE

**TEMOCAPRIL** 

TEMOCAPRIL HYDROCHLORIDE

**IMIDAPRIL** 

IMIDAPRIL HYDROCHLORIDE

MOEXIPRIL

MOEXIPRIL HYDROCHLORIDE

UDRAMIL

**ELIDIUR** 

LEXXEL

TECZEM /01366001/

VERACAPT

LASITACE

DELAPRIDE

PRIMOX PLUS

**UNIMAX** 

**BI PREDONIUM** 

**BENAZEPRILAT** 

**PENTOPRIL** 

IDRAPRIL

**MOVELTIPRIL** 

CERONAPRIL

TRANDOLAPRILAT

UTIBAPRIL

ZABICIPRIL





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


LIBENZAPRIL

**DINAPRES** 

OCADRIK /01507301/

ENEAS

CARACE PLUS /01613901/

AMLODIPINE W/BENAZEPRIL

AMLODIPINE BESYLATE W/BENAZEPRIL ALENDRONATE SODIUM W/QUINAPRIL

HYDROCHLORIDE

SINERGEN AMLOPRES L LORAM-H ENZIX

LOTRIX /03460001/

ARBITACE

ORAS /03528201/

TERAM
NAPRIX A
ACEDIP
M 100240
VASCORIDE
CARDIO-PRES D
CARSIPRIL D
RAMICAR D
CVPILL

NORMATEN /06267401/

ATOCOR-R
MODLIP-CAD
OLMY-R
ADPACE
BIFRIL PLUS
PERINDO COMBI
COVERAM

PRETERAX ARGININE

ZESTORETIC

INDAPAMIDE W/PERINDOPRIL

HYDROCHLOROTHIAZIDE W/QUINAPRIL FOSINOPRIL W/HYDROCHLOROTHIAZIDE ENAP-HL /06436201/

CAPTOPRIL W/ENALAPRIL

DIRONORM POLYCAP ZOPRANOL PLUS





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


AMLODIPINE MALEATE W/BENAZEPRIL

**HYDROCHLORIDE** 

AMTAS PRP

CILAZAPRIL MONOHYDRATE W/HYDROCHLOROTHIAZIDE

GEMOPATRILAT

HYDROCHLOROTHIAZIDE W/MOEXIPRIL

FASIDOTRIL UTIBAPRILAT MOEXIPRILAT

MOEXIPRILAT HYDROCHLORIDE

**OMAPATRILAT** 

AMLODIPINE W/BENAZEPRIL HYDROCHLORIDE

BENAZEPRIL W/HYDROCHLOROTHIAZIDE

VIVACE /06864501/

CAPTRAL ASA RAMEY D STARPRESS R DILVAS AM R PRIL AM VALZAAR R

TERAM H METPURE AR

PERINDOPRIL ARG/AMLODIPINE FISHER

LOTRIAL VAS

**ENALAPRIL W/NITRENDIPINE** 

SINCRONIUM /07912401/

COROVAL B ZANERIL

ENALAPRIL W/LERCANIDIPINE

RAMITORVA METOZ R MET XL R RAMI ASOMEX

PERINDOPRIL TOSILATE/ INDAPAMIDE

METOPROLOL W/RAMIPRIL

SAMPATRILAT

AMLODIPINE W/INDAPAMIDE/PERINDOPRIL

GLIMEPIRIDE W/METFORMIN HYDROCHLORIDE/RAMIPRI ATORVASTATIN CALCIUM W/GLIMEPIRIDE//08698201/ AMLODIPINE BESILATE W/INDAPAMIDE/PE/08715301/

AMLODIPINE BESILATE W/PERINDOPRIL TOSILATE





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

| | AMLODIPINE BESILATE |
|-------------------|--------------------------------------|
| | W/INDAPAMIDE/PE/08717501/ |
| | AMLODIPINE W/LISINOPRIL/ROSUVASTATIN |
| | TEMOCAPRILAT |
| | INDAPAMIDE HEMIHYDRATE W/PERINDOPRIL |
| | ARGININE |
| | ACE INHIBITORS, PLAIN |
| | ACE INHIBITORS, COMBINATIONS |
| | ACE INHIBITORS AND CALCIUM CHANNEL |
| | BLOCKERS |
| | ACE INHIBITORS |
| Angiotensin | LOSARTAN |
| _ | LOSARTAN POTASSIUM |
| receptor blockers | HYZAAR |
| | TASOSARTAN |
| | SAPRISARTAN |
| | SAPRISARTAN POTASSIUM |
| | VALSARTAN |
| | IRBESARTAN |
| | IRBESARTAN HYDROCHLORIDE |
| | CO-DIOVAN |
| | EPROSARTAN |
| | EPROSARTAN MESILATE |
| | CANDESARTAN |
| | CANDESARTAN CILEXETIL |
| | KARVEA HCT |
| | BLOPRESS PLUS |
| | TELMISARTAN |
| | HYDROCHLOROTHIAZIDE W/LOSARTAN |
| | AMLODIPINE W/VALSARTAN |
| | OLMESARTAN |
| | OLMESARTAN MEDOXOMIL |
| | BENICAR HCT |
| | CANDESARTAN W/HYDROCHLOROTHIAZIDE |
| | LOTAR /02225901/ |
| | DIOVAN AMLO |
| | LORAM-H |
| | NUSAR-ATN |
| | ARBITACE |
| | ORAS /03528201/ |
| | TERAM |
| | DIOCOMB SI |
| | AZOR /06230801/ |
| | AMLOZAAR-H |
| | TWYNSTA |
| | TELSAR-A |
| | DIOVAN TRIPLE |
| | OLMY-R |
| | LOSAR BETA-H |
| | ADPACE |





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


**VALTURNA** 

**EMBUSARTAN** 

**PRITORPLUS** 

**EMESTAR PLUS** 

NIFEDIPINE W/TELMISARTAN

HYDROCHLOROTHIAZIDE W/OLMESARTAN

COZAAR XQ PLEOTOR T

BENITEC A /06541301/

OLMESAFE AM CANDESAR A **TRIBENZOR** ATACAND DUO **ABITESARTAN** 

**RIPISARTAN** 

**AZILSARTAN** 

AZILSARTAN MEDOXOMIL AZILSARTAN KAMEDOXOMIL

**POMISARTAN PRATOSARTAN** FENSARTAN UNIMAX

OLSAR M

AZELNIDIPINE W/OLMESARTAN MEDOXOMIL

OLMAT AMH **AMLODIPINE** 

W/HYDROCHLOROTHIAZIDE/VALSARTAN

CO IRABEL CILACAR T INDITEL D ZIVAST L VALZAAR R

NEBICARD V TERAM H

**RASOTAN BETA TELISTA MT** 

**TELMICHEK AH EDARBYCLOR FIMASARTAN** 

FIMASARTAN POTASSIUM TRIHYDRATE

**TELROSE** CTD L ARBITEL MT

TAH

**APROVASC** 

AMLODIPINE W/OLMESARTAN

**ERITEL CH OLMESAT ID** 

ALISKIREN W/VALSARTAN

METOZ L

METOPROLOL W/TELMISARTAN





Clinical Study Report: 20140254 Primary Analysis


Product: AMG 334

Statistical Analysis Plan: 20140254


ASOMEX TM OLMESAR AV

ASOMEX LTH

IRBESARTAN W/TRICHLORMETHIAZIDE FIMASARTAN POTASSIUM TRIHYDRATE

W/HYDROCHLORO

LERCANIDIPINE HYDROCHLORIDE W/VALSARTAN

LEVAMLODIPINE BESILATE W/VALSARTAN AMLODIPINE W/CHLORTALIDONE/LOSARTAN

**POTASSIUM** 

CHLORTALIDONE W/OLMESARTAN MEDOXOMIL CILNIDIPINE W/OLMESARTAN MEDOXOMIL AMLODIPINE OROTATE W/VALSARTAN

AMLODIPINE MESILATE

W/HYDROCHLOROTHIAZIDE/VAL

ATORVASTATIN CALCIUM W/IRBESARTAN

AMLODIPINE W/CHLORTALIDONE/OLMESARTAN

MEDOXOM

AMLODIPINE W/CHLORTALIDONE/TELMISARTAN OLMESARTAN MEDOXOMIL W/ROSUVASTATIN CALCIUM

CILNIDIPINE W/VALSARTAN

ROSUVASTATIN CALCIUM W/VALSARTAN AMLODIPINE BESILATE W/AZILSARTAN AMLODIPINE BESILATE W/CANDESARTAN

CILEXETIL/H

AMLODIPINE ADIPATE W/VALSARTAN

CHLORTALIDONE W/CILNIDIPINE/TELMISARTAN

AMLODIPINE OROTATE W/OLMESARTAN

**MEDOXOMIL** 

SACUBITRIL W/VALSARTAN

ANGIOTENSIN II ANTAGONISTS, PLAIN

ANGIOTENSIN II ANTAGONISTS, COMBINATIONS ANGIOTENSIN II ANTAGONISTS AND CALCIUM

CHANNE



